CLINICAL TRIAL: NCT06147479
Title: Cognitive Stimulation in Activities of Daily Living for Individuals Living With Mild-to-Moderate Dementia (CS-ADL): a Pilot Randomised Controlled Trial
Brief Title: Cognitive Stimulation in Daily Activities for People Living With Early to Middle Stage Dementia
Acronym: CS-ADL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National University of Ireland, Galway, Ireland (Other)
Responsible Party: Principal Investigator, Simone Ryan, Principal Investigator; Occupational Therapist, National University of Ireland, Galway, Ireland
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: REC/23/042
Record Dates: First submitted 2023-11-15; First posted 2023-11-27 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Dementia; Dementia, Mild; Dementia Moderate
Keywords: Cognitive stimulation; Occupational therapy; randomised controlled trial; Activities of daily living; ADL
MeSH Terms: conditions — Dementia; Lymphoma, Follicular | interventions — Activities of Daily Living

STUDY DESIGN:
Intervention Model Description: This will be a multi-center, parallel, single-blind, randomized trial of CS-ADL versus treatment as usual for people with mild-to-moderate dementia.
Who Masked: Outcomes Assessor
Masking Description: The outcomes assessor will be blinded to group allocation where possible.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CS-ADL (Experimental): CS-ADL is a multi-component cognitive stimulation program that aims to enhance performance of activities of daily living (ADL) for people living with mild-to-moderate dementia.
  Interventions: Behavioral: CS-ADL (Cognitive stimulation in Activities of Daily Living)
- Treatment as Usual (TAU) (No Intervention): The control group continue to receive their usual care. This may differ between individuals, but may include physiotherapy, occupational therapy, nursing, medication or attendance at a day-care centre/day hospital. This treatment is decided by their healthcare provider who is external to the research team. It is possible that 'TAU' for some individuals dictates no treatment.

INTERVENTIONS:
Behavioral: CS-ADL (Cognitive stimulation in Activities of Daily Living) — CS-ADL sessions are delivered once weekly, for seven weeks. Sessions last approximately 2 hours. Sessions are themed around domains of everyday activities, for example 'Morning routine', ' Domestic Activities', 'Leisure'. Activities in each session follow this theme. A typical session begins with introductions, reality orientation, a group song and discussion of the news of the week. This is followed by a physical activity/game and ADL-focused cognitive stimulation activities. These activities include the identification and categorization of everyday items, discussion, reminiscence, planning and sequencing of ADLs and the completion of everyday writing/calculation tasks. This is followed by practice of an ADL. Examples of activities include making a breakfast, a simple gardening activity or sorting laundry. The session then ends with a summary and repeat of the group song, and a plan for the next session.
  Arms: CS-ADL

SUMMARY:
The goal of this study is to test the effect of CS-ADL is on people living with early to middle stage dementia. The study also aims to evaluate the feasibility of conducting larger-scale research of CS-ADL.

The main questions it aims to answer are:

* What is the effect of CS-ADL on the ability of people with early to middle stage dementia to carry out their everyday activities?
* What is the effect of CS-ADL on the memory, mood, communication, and quality of life of people living with early to middle stage dementia? What is the feasibility of conducting large-scale research of CS-ADL?

Participants will take part in a group program that lasts 7 weeks, with one session per week, lasting two hours. Participants will take part in rewarding and stimulating activities, for example discussion, reminiscence, music, and practical activities such as baking, cooking, gardening. Participants will be asked to complete a variety of questionnaires before and after taking part in the group.

Researchers will compare a group receiving CS-ADL to a group receiving their usual care, to explore whether CS-ADL works well in comparison to typical treatment provided by the health services.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have a formal diagnosis of major neurocognitive disorder (dementia) as per the DSM-V criteria.
* Participants must have a mild-to-moderate cognitive impairment as classified by the Montreal Cognitive Assessment (MoCA).
* Participants must have some ability to communicate and understand communication, determined by a score of 1 or 0 on questions 12 and 13 of the Clifton Assessment Procedures for the Elderly-Behaviour Rating Scale.
* Participants must be able to see and hear well enough to participate in the group.

Exclusion Criteria:

* Individuals with severe dementia, i.e., an MMSE<10, will be excluded as most CS interventions are not applicable for those with severe cognitive impairment.
* Participants will be excluded if they have significant uncontrolled disruptive behaviours.
* Premorbid diagnosis of a learning disability.
* A significant physical illness/disability that may affect participation during intervention sessions or assessments.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2023-11-03 (Actual); Primary Completion 2024-06-21 (Actual); Study Completion 2024-06-21 (Actual)

PRIMARY OUTCOMES:
Change from baseline in the performance of activities of daily living (ADL) of participants | This will be administered at baseline (week 0), and post-intervention (week 8).
  ADL performance will be measured using the Alzheimer's Disease Cooperative Study-Activities of Daily Living (ADCS-ADL) scale. This scale was designed for the assessment of ADL outcomes for individuals with Alzheimer's disease in clinical trials. The scale consists of 23 items that includes 6 BADL and 17 IADL outcomes, scored on a range from 0 (patient does not perform the activity), to the highest score (patient is independent in the activity). The scale is administered with caregivers who are asked to rate the degree to which their care-recipient performs each item in the last four weeks. The ADCS-ADL has been identified to be a reliable and valid instrument, with high internal consistency and sensitivity to functional changes in individuals with mild-to-moderate dementia.

SECONDARY OUTCOMES:
Change from baseline in the global cognitive functioning of participants | This will be administered at baseline (week 0), and post-intervention (week 8).
  This outcome will be measured using Montreal Cognitive Assessment (Blind). The MoCA-Blind is scored on a scale of 22 points as visual elements are excluded. Specificity remains on par with the original MoCA. Scores from the MoCA-Blind are converted to align with the scores of the original MoCA using the following equation (result multiplied by 30) divided by 22. The interpretation ranges of scores are as follows: a score of 18-25 points indicates mild cognitive impairment; 10-17 points indicates moderate cognitive impairment; and fewer than 10 points indicates severe cognitive impairment. Scores ranging from 26 to 30 are considered as normal.
Change from baseline in cognition of participants | This will be administered at baseline (week 0), and post-intervention (week 8).
  Cognition will be assessed using the Repeatable Battery for Assessment of Neuropsychological Status (RBANS). The RBANS is a commonly used brief battery of cognitive function for individuals with dementia. This battery consists of 12 subtests which assess five cognitive domains: immediate memory, visuospatial-constructional ability, language and delayed memory. This battery has demonstrated good reliability and adequate validity indicators. Scores on the RBANS can range from 40 to 160, with a lower score indicating more severe cognitive impairment.
Change from baseline in communication ability of participants | This will be administered at baseline (week 0), and post-intervention (week 8).
  Communication ability will be assessed using the Holden Communication Scale (HCS). This scale includes 12 items assessing the domains of conversation, awareness, humour, and responsiveness. Each items contains five response options ranging from 0 to 4. Total scores can range from 0 to 48 with higher scores indicating more communication difficulties. The HCS was initially developed to assess communication outcomes in reality orientation and reminiscence programs and has demonstrated good reliability and validity for use with PLwD. While there are limitations to reliability and validity data outside of the original development of the tool, the HCS has been used in various CS studies to assess communication.
Change from baseline in quality of life of participants | This will be administered at baseline (week 0), and post-intervention (week 8).
  QOL will be assessed using the Quality of Life-Alzheimer's Disease Scale (QOL-AD). This scale consists of 13 items spanning the domains of physical health, energy, mood, living situation, memory, family, marriage, friends, chores, fun, money, self, and life as a whole. Response options include 1 (poor), 2 (fair), 3 (good) and 4 (excellent), with total scores ranging from 13-52. Higher scores indicate better quality of life. Assessment is delivered through an interview format and separate ratings are obtained from the participant themselves and the caregiver. Higher scores indicate a better quality of life. The QOL-AD has demonstrated good reliability and internal consistency and has been found to detect improvements in QOL in previous CS studies.
Change from baseline in neuropsychiatric symptoms of participants | This will be administered at baseline (week 0), and post-intervention (week 8).
  Mood will be assessed through the presence of neuropsychiatric symptoms as measured by the Neuropsychiatric Inventory Questionnaire (NPI-Q), a version of the Neuropsychiatric Inventory (NPI). The NPI-Q is a caregiver-based questionnaire that measures the presence and severity of 12 neuropsychiatric symptoms in PLwD, including delusions, hallucinations, apathy, disinhibition, and agitation/aggression. The severity scale runs from 1 to 3 points (1=mild, 2=moderate, 3=severe). The questionnaire also measures the respective level of caregiver distress associated with each symptom, with the scale running from 0 to 5 points (0=no distress, 5=extreme distress). The minimum score is 0 and the maximum score is 36, with higher scores indicating increased presence of neuropsychiatric symptoms. The scale is widely used in research, has demonstrated acceptable levels of internal consistency.

OTHER OUTCOMES:
Occupational performance within a group setting | This will be rated by the group facilitators following each session (week 1,2,3,4,5,6,7).
  Occupational performance within a group setting will be measured after each session using the Occupational Therapy Task Observation Scale (OTTOS). The OTTOS contains two parts, with 10 items for evaluation of specific task functions and 5 items for rating general behavior. The maximum total scores for both task behavior and general behavior are 100, with the minimum being 0 for both. Higher scores indicate greater functional behavior, with lower scores indicating dysfunctional behavior. The reliability and validity of the OTTOS has been demonstrateD.

CONTACTS AND LOCATIONS:
Overall Officials: Simone Ryan, BSc, Principal Investigator — University of Galway
Locations (1):
- University of Galway, Galway, Connacht, Ireland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ryan SM, Brady O. Cognitive stimulation in activities of daily living for individuals with mild-to-moderate dementia (CS-ADL): Study protocol for a randomised controlled trial. PLoS One. 2024 Sep 3;19(9):e0309337. doi: 10.1371/journal.pone.0309337. eCollection 2024. PMID 39226247